CLINICAL TRIAL: NCT00604578
Title: A Randomized, Placebo-Controlled, Double-Blind Pilot Study of Pioglitazone Hydrochloride in Allergic Asthma
Brief Title: Pioglitazone Hydrochloride (Actos(Registered Trademark)) to Treat Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Stewart J. Levine, M.D./National Heart, Lung, and Blood Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080047; 08-H-0047
Record Dates: First submitted 2008-01-08; First posted 2008-01-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-30

CONDITIONS: Asthma; Airway Inflammation; Airflow Obstruction; Airway Hyperactivity
Keywords: Pioglitazone; Asthma; Peroxisome Proliferator-Advanced Receptor Gamma; Airflow Obstruction; Airway Inflammation
MeSH Terms: conditions — Asthma | interventions — Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone Hydrochloride

SUMMARY:
This study will test whether pioglitazone hydrochloride (Actos (Registered Trademark) Registered Trademark) is effective for treating patients with asthma who do not respond to standard therapy. Experiments have shown that this drug, which is used to treat patients with diabetes, may be effective for treating asthma.

People between 18 and 75 years of age who have had asthma for at least a1 year and whose symptoms are not well controlled with high doses of inhaled corticosteroids with or without long-acting bronchodilators may be eligible for this study. Candidates are screened with breathing tests, an allergy skin test, chest x-ray, electrocardiogram (ECG), echocardiogram (ultrasound test of the heart), blood tests, and DEXA scan (an x-ray to measure bone thickness) to make sure they are eligible for the study.

Then, participants undergo tests and procedures in the following study phases:

Phase 1

Participants are given a device to measure and record their lung function and asthma symptoms at home each morning and night for 4 weeks before starting the study medication. Lung function is also measured at clinic visits before and after inhaling a bronchodilator medicine. Before starting the study medication, participants have a sputum induction (sputum collection test). For this test, the participants inhale a salt-water mist and are asked to collect sputum into a plastic cup.

Phase II

Participants are randomly selected to receive either pioglitazone hydrochloride or placebo (a look-alike pill with no active ingredient) once a day for 10 weeks. They return to the clinic after 2 weeks to repeat the tests done in Phase 1 and to monitor any reactions to the study drug or placebo. If there are no problems, the amount of medication is increased once, and then they return for follow-up evaluations every 2 weeks for 8 weeks. Pulmonary function tests, sputum collection and DEXA scan are repeated after 10 weeks on medication.

Phase III

Patients return for follow-up 1 month after stopping the medication or placebo to monitor their asthma.

...

DETAILED DESCRIPTION:
New therapies are needed for patients with asthma who are suboptimally controlled by standard measures. Pioglitazone hydrochloride (Actos [R]) is a highly selective and potent agonist for the peroxisome proliferator-activated receptor-gamma (PPAR gamma). Studies in murine models of allergic asthma have shown that PPAR gamma-agonists down-regulate allergen-mediated airway inflammation and airway hyperresponsiveness. This protocol is a randomized, placebo-controlled, double-blind, parallel-group (phase II) pilot study of the efficacy and safety of pioglitazone for the treatment of patients with allergic asthma and reversible airflow obstruction who are persistently symptomatic despite therapy with high doses of inhaled corticosteroids with or without long-acting Beta 2-agonists. The primary end-point for this study will be the change in airflow obstruction, as measured by the post-bronchodilator FEV1. Secondary end-points will include indices of airway inflammation, airflow obstruction, airway hyperreactivity, and asthma symptoms.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be between 18 and 75 years of age, male or female, with a diagnosis of asthma for at least one year.

Patients must have reversible airflow obstruction as defined by a positive methacholine bronchoprovocation challenge or a positive response to inhaled bronchodilators.

Patients must be treated with EPR-3 Step 5 therapy (high dose (great than or equal to 440 ucg/day) fluticasone inhaler or equivalent dose of another inhaled corticosteroid) with or without an inhaled long-acting beta-2-agonist) for at least 3 months.

Patients must meet the EPR-3 criteria for not well controlled asthma. The EPR-3 definition for not well controlled asthma includes any of the following features in a week (unless otherwise indicated): daytime asthma symptoms great than 2 days/week, limitation of activities, nocturnal symptoms or awakening greater than 2 times/month, need for reliever/rescue treatment greater than 2 days/week, PEF or FEV(1) less than 80% predicted.

Pre-bronchodilator FEV(1) greater than or equal to 55% of predicted and post-bronchodilator FEV(1) greater than or equal to 60% of predicted.

During the 6 weeks prior to enrollment, patients should have stable asthma as defined by the absence of unscheduled health care visits for asthma care and unchanged use of asthma maintenance therapy. Additional criteria for disease stability include the absence of hospitalization for asthma or the need for a course of oral corticosteroids during the preceding 3 months.

Research subjects must have a positive skin test to a common aeroallergen, such as dust mite, cat, short ragweed, cockroach, or grass or a prior history of severe allergy or anaphylaxis.

Chest radiograph without evidence of pulmonary disease, other than asthma.

Left ventricular ejection fraction greater than or equal to 50% by echocardiogram.

For women of childbearing potential, negative pregnancy test within 2 weeks prior to study and willingness to adhere to reliable birth control methods during the study.

Subjects with a history of dermatologic cancers may be included if they have been cancer-free for at least 5 years prior to enrollment.

EXCLUSION CRITERIA:

A known history of hypersensitivity to pioglitazone.

Maintenance asthma therapy with oral corticosteroids, xolair (anti-IgE), methotrexate, cytoxan, gold salts, or cyclosporine.

Cigarette smoking within the past 3 months or a prior history of greater than 10 cumulative pack-years.

Viral or bacterial upper respiratory tract infection within 6 weeks prior to the screening visit.

Investigational therapy for any indication within 1 month prior to the screening visit.

History of lung disease other than asthma (i.e., COPD, sarcoidosis).

History of diabetes mellitus, insulin secreting tumor, or symptomatic hypoglycemia.

HIV or other known immunodeficiency.

History of congestive heart failure.

Preexisting edema (2 plus or greater).

Hemoglobin less than 12 gm/dl for males and less than 11 gm/dl for females.

History of liver disease or abnormal liver function tests greater than 2 times upper limit of normal.

History of inflammatory bowel disease.

History of cancer (other than dermatologic cancer).

History of drug or alcohol abuse.

Use of the following medications, which can interact with pioglitazone:

Gemfibrizol (Lopid)

Atazanivir (Reyataz)

Ritonavir (Norvir)

Rifampin (Rifampicin)

Carbamzepine (Tegretol)

Phenobarbital (Luminal)

Phenytoin (Dilantin)

Rifapentine (Priftin)

Secobarbital (Seconal)

Amiodarone (Cordarone, Pacerone)

Palitaxel (Taxol)

Replaglinide (Prandine)

Ketoconazole (Nizoral)

Atorvastatin (Lipitor(Registered Trademark))

Nifedipine ER (Adalat CC)

Any condition that, in the investigator's opinion, places the patient at undue risk for complications from pioglitazone therapy.

Dexa bone scan (T score below -1 SD).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01-04; Primary Completion 2009-10-30 (Estimated); Study Completion 2009-10-30 (Estimated)

PRIMARY OUTCOMES:
The change in post-bronchodilator FEV1. | 10 weeks

SECONDARY OUTCOMES:
Airway inflammation, Airflow Obstruction, Airway Hyperreactivity, Asthma Symptoms, Rate of mild exacerbation, Rate of severe exacerbation, Asthma Quality-of-life, Blood Eosinophil Counts, Serum IgE and Exhaled Nitric Oxide Levels. | 10 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Background] Wenzel SE. Asthma: defining of the persistent adult phenotypes. Lancet. 2006 Aug 26;368(9537):804-13. doi: 10.1016/S0140-6736(06)69290-8. PMID 16935691
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] Strunk RC, Bloomberg GR. Omalizumab for asthma. N Engl J Med. 2006 Jun 22;354(25):2689-95. doi: 10.1056/NEJMct055184. No abstract available. PMID 16790701